CLINICAL TRIAL: NCT06305598
Title: Bipolar Androgen Therapy in Metastatic Castration-Resistant Prostate Cancer (mCRPC)
Brief Title: Bipolar Androgen Therapy to Restore Sensitivity to Androgen Deprivation Therapy for Patients With Metastatic Castration Resistant Prostate Cancer
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Roswell Park Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: I-3298823; NCI-2024-01390 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); I-3298823 (Other: Roswell Park Cancer Institute)
Record Dates: First submitted 2024-03-05; First posted 2024-03-12 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Castration-Resistant Prostate Carcinoma; Metastatic Prostate Carcinoma; Stage IVB Prostate Cancer AJCC v8
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Biopsy; Leuprolide; luprolide acetate gel depot; Magnetic Resonance Spectroscopy; testosterone 17 beta-cypionate; Testosterone Propionate; Methyltestosterone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Treatment (Bipolar androgen therapy) (Experimental): Patients receive testosterone IM on day 1 of each cycle. Cycles repeat every 28 days for 3 cycles in the absence of disease progression or unacceptable toxicity. Patients also continue to receive standard of care leuprolide acetate SC per their standard schedule. Patients undergo CT scan, bone scan and may undergo MRI and tumor biopsy throughout the study.
  Interventions: Procedure: Biopsy; Procedure: Bone Scan; Procedure: Computed Tomography; Drug: Leuprolide Acetate; Procedure: Magnetic Resonance Imaging; Other: Survey Administration; Drug: Testosterone Cypionate

INTERVENTIONS:
Procedure: Biopsy — Undergo biopsy
  Other Names: BIOPSY_TYPE; Bx
Procedure: Bone Scan — Undergo bone scan
  Other Names: Bone Scintigraphy
Procedure: Computed Tomography — Undergo CT scan
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; tomography
Drug: Leuprolide Acetate — Given SC
  Other Names: A-43818; Abbott 43818; Abbott-43818; Carcinil; Depo-Eligard; Eligard; Enanton; Enantone; Enantone-Gyn; Ginecrin; LEUP; Leuplin; Leuprorelin Acetate; Lucrin; Lucrin Depot; Luprodex Depot; Lupron; Lupron Depot; Lupron Depot-3 Month; Lupron Depot-4 Month; Lupron Depot-Ped; Lutrate; Procren; Procrin; Prostap; TAP-144; Trenantone; Uno-Enantone; Viadur
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Other: Survey Administration — Ancillary studies
Drug: Testosterone Cypionate — Given IM
  Other Names: depAndro; Depo-Testosterone; Depotest; Depovirin; Pertestis; Virilon

SUMMARY:
This phase I trial tests the change in androgen receptor sensitivity, side effects and effectiveness of bipolar androgen therapy, using testosterone, in patients with castration resistant prostate cancer that has spread to other places is the body (metastatic). Bipolar androgen therapy is the regulation of testosterone between castration levels (lower than what would be normally present) and supraphysiological levels (amounts greater than normally found in the body). This may suppress cancer cell growth, which reduces prostate-specific antigen (PSA) levels and may delay cancer progression.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the influence of bipolar androgen therapy (BAT) on androgen receptor (AR) activity in patients with metastatic castration-resistant prostate cancer (mCRPC).

SECONDARY OBJECTIVES:

* To determine the clinical efficacy and safety of BAT in patients with mCRPC.
* To determine the change in fatigue and quality of life in patients receiving BAT.

OUTLINE:

Patients receive testosterone intramuscularly (IM) on day 1 of each cycle. Cycles repeat every 28 days for 3 cycles in the absence of disease progression or unacceptable toxicity. Patients also continue to receive standard of care leuprolide acetate subcutaneously (SC) per their standard schedule. Patients undergo computed tomography (CT) scan, bone scan and may undergo magnetic resonance imaging and tumor biopsy throughout the study.

After completion of study treatment, patients follow up at 30 days and every 3 months for up to 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years of age
* Have an Eastern Cooperative Oncology Group (ECOG) performance status of ≤ 2
* Histologically confirmed carcinoma of the prostate
* Progressing on continuous androgen ablative therapy (either surgical castration or LHRH agonist)
* Documented castrate level of blood testosterone (< 50 ng/dL)
* Patients must have progressed on prior treatment with at least one Androgen Receptor Signaling Inhibitors (ARSI) (by prostate specific antigen [PSA] criteria or radiographically)
* Have biopsiable disease (a fresh biopsy is not required at baseline if adequate archival tissue is available)
* Absolute neutrophil count: ≥1,200/µL
* Platelets: ≥ 100,000/µL
* Total bilirubin: ≤ 1.2 x institutional upper limit of normal (ULN)
* Aspartate aminotransferase (AST)(serum glutamic oxaloacetic transaminase [SGOT])/ Alanine aminotransferase (ALT) (serum glutamic pyruvic transaminase [SGPT]): ≤ 3 × institutional ULN
* Creatinine clearance (CrCl) > 50 mL/min (Cockcroft-Gault equation)
* Have measurable disease per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 criteria present
* Participants of child-bearing potential must agree to use adequate contraceptive methods (e.g., hormonal or barrier method of birth control; abstinence) prior to study entry. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately
* Participant must understand the investigational nature of this study and sign an Independent Ethics Committee/Institutional Review Board approved written informed consent form prior to receiving any study related procedure

Exclusion Criteria:

* Participants who have had chemotherapy or radiotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier
* Participants with known brain metastases should be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events
* Greater than 5 sites of visceral disease in lung or liver (nonspecific lung nodules ≤ 1 cm in diameter is permitted)
* Evidence of disease in sites or extent that, in the opinion of the investigator, would put the patient at risk from therapy with testosterone (e.g., femoral metastases with concern over fracture risk, spinal metastases with concern over spinal cord compression, lymph node disease with concern for ureteral obstruction)
* Active uncontrolled infection, including known history of acquired immunodeficiency syndrome (AIDS) or hepatitis B or C
* Any psychological, familial, sociological, or geographical condition that could potentially interfere with compliance with the study protocol and follow-up schedule
* Prior history of a thromboembolic event within the last 12 months and not currently on systemic anticoagulation
* Hematocrit > 50%, untreated severe obstructive sleep apnea, uncontrolled or poorly controlled heart failure (per Endocrine Society Clinical Practice Guidelines)
* Evidence of serious and/or unstable pre-existing medical, psychiatric, or other condition (including laboratory abnormalities) that could interfere with patient safety or provision of informed consent to participate in this study
* Known allergy to testosterone cypionate or any of its excipients
* Unwilling or unable to follow protocol requirements
* Any condition which in the Investigator's opinion deems the participant an unsuitable candidate to receive study drug

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Estimated)
Dates: Start 2024-12-19 (Actual); Primary Completion 2026-12-15 (Estimated); Study Completion 2027-12-15 (Estimated)

PRIMARY OUTCOMES:
Androgen receptor (AR) activity | Up to 2 years after end of treatment/progression
  Assessed with spatial transcriptomic profiling using the well-validated Nelson 10 genes signature AR score. Will be summarized by timepoint using the mean and standard deviation, and graphically using dot-plots. The mean pre/post-intervention levels will be compared using a one-sided paired t-test (expected increase); with the effect summarized using the mean difference and fold change.

SECONDARY OUTCOMES:
Incidence of adverse events | Up to 30 days after end of treatment or progression
  Using the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 5.0.
Incidence of serious adverse events | Up to 30 days after end of treatment or progression
  Using the NCI CTCAE version 5.0.
Prostate specific antigen (PSA) 50 | Up to 2 years after end of treatment/progression
  Defined as the proportion of patients with a >=50% reduction in PSA from the maximal PSA level achieved during the treatment. Will be summarized using frequencies and relative frequencies.
Measurable disease response | Up to 2 years after end of treatment/progression
  Will be summarized using frequencies and relative frequencies.
Progression free survival | From day 1 of treatment to the date when the first site of disease is found to progress, assessed up to 2 years after end of treatment/progression
  Will be summarized using standard Kaplan-Meier methods, where the medians will be estimated with 95% confidence intervals (CIs).
Overall survival | From the time of initiation of treatment until death from any cause, assessed up to 2 years after end of treatment/progression
  Will be summarized using standard Kaplan-Meier methods, where the medians will be estimated with 95% CIs.
Assess Quality of life | Up to 2 years after end of treatment/progression
  Using the FACIT-F.he FACIT-F is a well-validated QOL instrument widely used for the assessment of cancer-related fatigue in clinical trials. It consists of 27 general QOL questions divided into 4 domains (physical, social, emotional, and functional), plus a 13-item fatigue sub-score. The patient rates the intensity of fatigue and its related symptoms on a scale of 0-4. The total score ranges between 0 and 52, with higher scores denoting less fatigue . Comparisons will be made between pre- and post-treatment using a paired t-test.
Assess Quality of Life | Up to 2 years after end of treatment/progression
  A self-reported 36 item survey (SF-36) of patient health where higher scores indicated better health related quality of life
Assess Fatigue | Up to 2 years after end of treatment/progression
  Using the FACIT-F (FACIT Fatigue Scale) the FACIT-F is a well-validated QOL instrument widely used for the assessment of cancer-related fatigue in clinical trials. It consists of 27 general QOL questions divided into 4 domains (physical, social, emotional, and functional), plus a 13-item fatigue sub-score. The patient rates the intensity of fatigue and its related symptoms on a scale of 0-4. The total score ranges between 0 and 52, with higher scores denoting less fatigue
Assess change in Fatigue | Up to 2 years after end of treatment/progression
  Assess changes in Fatigue using the SF-36 (Short Form Health Survey) A self reported 36 item survey where lower scores indicate greater fatigue.

CONTACTS AND LOCATIONS:
Overall Officials: Gurkamal S Chatta, Principal Investigator — Roswell Park Cancer Institute
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States